CLINICAL TRIAL: NCT06894810
Title: A Double Blind Randomised Controlled Trial of a Paediatric Fertility Preservation Decision Aid in Parents and Adolescents and Young Adults (CAYA) Cancer Survivors
Brief Title: Investigating the Efficacy of a Paediatric Fertility Preservation Decision Aid in Parents and Adolescents and Young Adults (CAYA) Cancer Survivors
Acronym: FOCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HREC 107901
Record Dates: First submitted 2025-02-20; First posted 2025-03-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-06

CONDITIONS: Unmet Fertility Information Needs
Keywords: Fertility preservation; Child Adolescent and Young Adults; Decision Aid; CAYA; Cancer Survivors
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid group (Active Comparator): Participants will have access to fertility preservation Decision Aid (DA) in addition to high-quality information (intervention group).
  Interventions: Other: Decision-aid
- CanTeen group (No Intervention): Participants will have access to high-quality information from CanTeen website (Control group).

INTERVENTIONS:
Other: Decision-aid — Decision Aids (DA) are evidence-based clinical tools developed for patients to supplement clinicians' discussions and facilitate difficult preference-sensitive decisions. They are the gold standard approach (recommended by the Australian Commission of Safety and Quality in Healthcare) to facilitate complex healthcare decisions where there is more than one reasonable choice and where patients may value benefits and risks differently.
  Arms: Decision aid group

SUMMARY:
The current standard of care for paediatric patients with cancer regarding preservation of their fertility (FP) is to provide high-quality information during the clinical consultation process. However, this approach depends on health provider knowledge and communication and has been shown to be sub-optimal in some situations. This impairs the critical decision-making of patients regarding fertility testing, utilization of gametes, and continuing payment of storage fees. The fertility preservation decision aid (FP DA) may lead to a greater understanding of their fertility status for participants. This knowledge may allow participants the opportunity to assess potential fertility issues prior to the end of their reproductive window, helping to minimize missed opportunities for parenthood.

This research study aims to assess the effectiveness of the use of the FP DA on unmet fertility information needs when it is provided in addition to high-quality information in parents of cancer survivors and CAYA cancer survivors compared to high-quality information alone.

DETAILED DESCRIPTION:
Medical advances over recent decades have increased the overall survival rates of children, adolescents and young adults diagnosed with cancer, with survival rates now exceeding 80%. The pressure points are not only at diagnosis - research has shown that cancer treatment can potentially affect fertility later in life. Survivorship is an important time for addressing the following issues: fertility status, reproductive monitoring, decisions about interval fertility preservation, ongoing tissue storage and utilization. Options to preserve fertility are possible. Decision Aids (DA) have been developed to provide patients and their families with the required information to make informed reproductive health decisions that align with their values. The prevalence of fertility information needs that are unmet remains high at around 40% amongst cancer survivors. Research evaluating the effectiveness of DAs in survivorship is lacking.

This is a parallel group double-blind randomised controlled trial for parents and Child Adolescent and Young Adults (CAYA) cancer survivors assessing the Fertility Preservation Decision Aid (FP DA) when provided in conjunction with high-quality information.

Eligible participants will be randomly allocated to either a control group receiving high-quality information or a treatment group that will receive the FP DA in addition to high-quality information. Participants will be blinded to their group allocation as they will be instructed to review information regarding fertility preservation without informing them of the type of information they are reviewing.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for both parents and survivors:

* Be able to communicate in English.
* Signed written informed consent form.

Inclusion Criteria for parents only:

• Parents/guardians of CAYA survivors who were ≤25 years (2) when diagnosed with cancer and have completed curative gonadotoxic treatment

Inclusion Criteria for survivors only

* CAYA cancer survivors aged 16 years or over who have completed curative gonadotoxic treatment.
* Participants can be on long-term adjuvant or endocrine therapy.
* Participants may have achieved a pregnancy or livebirth.

Exclusion Criteria:

Exclusion Criteria for both parents and survivors:

* CAYA patients currently undergoing cancer treatment and their parents/guardians.
* CAYA patients who are palliative and their parents/guardians
* A family member already in the study.

Exclusion Criteria for survivors only:

• Minors who are not deemed to be mature minors as per protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Unmet information needs as measured by the Unmet Information Needs Scale within 8 weeks of randomisation | within 8 weeks from randomisation
  Unmet information needs will be measured within 8 weeks post-randomisation using the Unmet Information Needs Scale. Items included in the questionnaire are: knowledge regarding fertility status, future parenthood goals, and information regarding fertility preservation procedures carried out at either the treatment or survivorship period. Needs are assessed on a 6-point scale, ranging from 0 to 5, with higher scores indicating greater unmet information needs.

SECONDARY OUTCOMES:
Change in unmet fertility information needs as measured by questionnaire at 6 months post-randomisation | 6 months post-randomisation
  Unmet fertility information needs will be measured at 6 months post-randomisation using the Unmet Information Needs Scale. Items included in the questionnaire are: knowledge regarding fertility status, future parenthood goals, and information regarding fertility preservation procedures carried out at either the treatment or survivorship period. Needs are assessed on a 6-point scale, ranging from 0 to 5, with higher scores indicating greater unmet information needs.
Change in fertility knowledge as measured using a purposively designed knowledge scale within 8 weeks of randomisation and at 6 months post-randomisation | within 8 weeks of randomisation, 6 months after randomisation
  Changes in fertility knowledge will be measured using a purposively designed knowledge scale within 8 weeks of randomisation and at 6 months after randomisation. The knowledge scale that ranges from 0 to 6, with higher values indicated better knowledge.
Change in decision making preparedness regarding fertility preservation measured by the Preparation for Decision Making Scale within 8 weeks of randomisation and at 6 months post-randomisation | within 8 weeks of randomisation, 6 months after randomisation
  Preparation for decision making will be measured by the utility of the information provided by participants using the Preparation for Decision Making Scale. The preparation for decision making scaling regarding fertility preservation comprises a 10 item scale with each answer scored 1 (not at all) to 5 (a great deal). The 10 items are summed and divided by 10. A higher score reflects greater preparation for decision making.
Change in decisional conflict as measured by the a validated decisional conflict scale within 8 weeks of randomisation and at 6 months post-randomisation | within 8 weeks and 6 months after randomisation
  Decisional conflict is defined as uncertainty around the decision to see a health professional for further advice about sexual and reproductive health and uncertainty around choices available to achieve parenthood. This will be measured using a validated decisional conflict scale. Scores range from 0 [feels extremely supported in decision making] to 100 [feels extremely unsupported in decision making].
Change in feasibility and acceptability of the information resources measured using a validated feasibility and acceptability scale within 8 weeks of randomisation and at 6 months post-randomisation | within 8 weeks of randomisation, 6 months after randomisation
  Feasibility and acceptability of using the information resources will be measured using a validated feasibility and acceptability scale. They are assessed on a 5-point scale, ranging from 1 to 5, with higher scores indicating greater feasibility and acceptability.
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- bounce rate | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- bounce rate will be collected using a first-party analytics provider (Mixpanel).
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- average session duration | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- average session duration will be collected using a first-party analytics provider (Mixpanel).
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- average time on pages | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- average time on pages will be collected using a first-party analytics provider (Mixpanel).
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- pages view per visit | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- total number of pages view across the website per visit will be collected using a first-party analytics provider (Mixpanel).
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- user behavior flow | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- user behavior flow will be collected using a first-party analytics provider (Mixpanel).
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- exit rate | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- exit rate will be collected using a first-party analytics provider (Mixpanel).
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- returning users | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- returning users will be collected using a first-party analytics provider (Mixpanel).
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- heatmap | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- heatmap will be collected using a first-party analytics provider (Mixpanel).
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- individual page rating | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- individual page rating will be collected using a first-party analytics provider (Mixpanel).
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- the proportion of values clarification exercises completed | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- the proportion of values clarification exercises completed will be collected using a first-party analytics provider (Mixpanel).
Change in Fertility Preservation Decision Aid (FP DA) usage analytic- the responses to the exercises | within 8 weeks of randomisation, 6 months after randomisation
  FP DA usage analytic- the responses to the exercises completed will be collected using a first-party analytics provider (Mixpanel).

OTHER OUTCOMES:
Changes in perceived usefulness of the information resources measured by a 5-item Decision Aid development scale at the time of diagnosis | within 8 weeks of randomisation, 6 months after randomisation
  A five-point scale, ranging from 0 to 4, adapted from a Decision Aid (DA) development study will be used to assess the perceived usefulness of the information resources as a decision-making tool and whether it would have been helpful at the time of diagnosis. The higher scores will indicate greater perceived usefulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Murdoch Children's Research Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
The current protocol states that data will not be shared. The protocol will be modified in due course to include data sharing and the record will be updated to reflect this.

REFERENCES:
- [Result] McDougall RJ, Gillam L, Delany C, Jayasinghe Y. Ethics of fertility preservation for prepubertal children: should clinicians offer procedures where efficacy is largely unproven? J Med Ethics. 2018 Jan;44(1):27-31. doi: 10.1136/medethics-2016-104042. Epub 2017 Oct 30. PMID 29084865
- [Result] Turcotte S, Guerrier M, Labrecque M, Robitaille H, Rivest LP, Hess B, Legare F. Dyadic validity of the Decisional Conflict Scale: common patient/physician measures of patient uncertainty were identified. J Clin Epidemiol. 2015 Aug;68(8):920-7. doi: 10.1016/j.jclinepi.2015.03.005. Epub 2015 Mar 21. PMID 25958108
- [Result] Lehmann V, Keim MC, Nahata L, Shultz EL, Klosky JL, Tuinman MA, Gerhardt CA. Fertility-related knowledge and reproductive goals in childhood cancer survivors: short communication. Hum Reprod. 2017 Nov 1;32(11):2250-2253. doi: 10.1093/humrep/dex297. PMID 29040512
- [Result] Benedict C, Stal J, Davis A, Zeidman A, Pons D, Schapira L, Diefenbach M, Ford JS. Greater fertility distress and avoidance relate to poorer decision making about family building after cancer among adolescent and young adult female survivors. Psychooncology. 2023 Oct;32(10):1606-1615. doi: 10.1002/pon.6212. Epub 2023 Sep 11. PMID 37695291